CLINICAL TRIAL: NCT00670033
Title: Comparison of Safety and IOP-Lowering Efficacy of Three Alternative Travoprost Formulations to Vehicle and TRAVATAN® in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Travoprost New Formulations in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-07-46
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-06

CONDITIONS: Ocular Hypertension; Open-angle Glaucoma
Keywords: IOP; Open-angle glaucoma; Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Travoprost new formulation (Experimental): Travoprost ophthalmic solution (new formulation), 1 of 3 dose levels, 1 drop in the study eye(s) once daily, at 8 PM, for 4 weeks
  Interventions: Drug: Travoprost ophthalmic solution (new formulation)
- TRAVATAN (Active Comparator): Travoprost ophthalmic solution 0.004%, 1 drop in the study eye(s) once daily, at 8 PM, for 4 weeks
  Interventions: Drug: Travoprost ophthalmic solution, 0.004%
- Vehicle (Placebo Comparator): Inactive ingredients, 1 drop in the study eye(s) once daily, at 8 PM, for 4 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Travoprost ophthalmic solution (new formulation)
  Arms: Travoprost new formulation
Drug: Travoprost ophthalmic solution, 0.004%
  Other Names: TRAVATAN®; TRAVATAN Z®
  Arms: TRAVATAN
Drug: Vehicle — Inactive ingredients used as a placebo
  Arms: Vehicle

SUMMARY:
The purpose of this study was to describe the safety and IOP-lowering efficacy of Travoprost New Formulations compared to TRAVATAN® and to vehicle in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy all informed consent requirements;
* Diagnosed with open-angle glaucoma or ocular hypertension;
* Able to discontinue use of all IOP-lowering medications for a minimum of 5 to 28 days prior to the Eligibility 1 Visit;
* IOP measurements in at least 1 eye as specified in protocol;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential if pregnant, breastfeeding, or not using highly effective birth control measures;
* Any form of glaucoma other than open-angle glaucoma;
* Severe central visual field loss in either eye;
* Chronic, recurrent or severe inflammatory eye disease;
* Clinically relevant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment, in the opinion of the Investigator;
* Best-corrected visual acuity (BCVA) worse than 0.60 logarithm of the miniminum angle of resolution (logMAR);
* Intraocular surgery within the past 6 months;
* Ocular laser surgery within the past 3 months;
* Any abnormality preventing reliable applanation tonometry;
* Severe illness or any other conditions which would make the patient, in the opinion of the Investigator, unsuitable for the study;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in intraocular pressure (IOP) | Baseline, Up to Week 4
  IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater amount of improvement.

SECONDARY OUTCOMES:
Mean intraocular pressure | Baseline, Up to Week 4
  IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Mean percent change from baseline in IOP | Baseline, Up to Week 4
  IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative percent change indicates a greater amount of improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, PhD, Study Director — Alcon Research